CLINICAL TRIAL: NCT01129232
Title: A Phase II-study (Therapeutic Exploratory) of GAD-alum in Newly Diagnosed Type-1 Diabetic Patients, With Focus One the Presence of Viruses at the Time of Diagnosis
Brief Title: Diabetes Virus Detection Project, Intervention With GAD-alum
Acronym: DiViD
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Complications to procedure
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Lars Krogvold, Assosciate professor, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2009/1907 (REK); 2008-002027-82 (EudraCT Number)
Record Dates: First submitted 2010-05-11; First posted 2010-05-24 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Diabetes, Type I; Enterovirus Infections; Autoimmunity
Keywords: insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Enterovirus Infections; Autoimmune Diseases; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GAD-alum (Experimental): GAD-alum administered at 0 and 1 months after inclusion
  Interventions: Drug: GAD-alum
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: GAD-alum — 20 µg of GAD-alum injected sc after the biopsy, and repeated after one month
  Other Names: Diamyd
  Arms: GAD-alum
Other: Placebo — Placebo injected after the biopsy and repeated after one month (similar to the GAD-alum-arm)
  Arms: Placebo

SUMMARY:
The purposes of this study are to test whether GAD vaccination can stop the progression of newly diagnosed type 1 diabetes, to describe the related immunological processes (insulitis) in pancreas and small intestines evolving the mechanism of the effect of GAD vaccination and finally try to detect viruses and virus receptors directly in the insulin producing beta cells of the pancreas in patients with newly diagnosed type-1 diabetes mellitus (T1D).

DETAILED DESCRIPTION:
The aetiology of type 1 diabetes is unknown. Both genetic and environmental factors seem to be important for the destruction of insulin producing beta cells in the pancreas. Increasing indirect evidences exist that picornaviruses may either directly or indirectly through autoimmune processes destroy beta cells. New sensitive assays have been developed to detect these viruses and to study the immunological processes, especially T-cell function. Microsurgical technology has been refined, now making pancreatic biopsies a safe procedure. This study focuses on advanced in depth studies of immunology and virology in pancreatic tissue and small intestine at an early stage of disease.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed classical type-1 diabetes
* Positive GAD antibodies
* Fasting C-peptide >0.1 mmol/l
* Insulin dosage >0.1 U/kg Bodyweight/day

Exclusion Criteria:

* Pregnancy
* Weaning
* Other chronic diseases than diabetes
* Any regular medication except oral contraceptives
* Psychiatric disturbances

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Intensity of insulitis in proportion to living, insulin-staining beta cells in pancreatic biopsies | 18 months after inclusion
Prevalence of virus infected islets in pancreatic biopsies | 18 months after inclusion
Intensity of insulitis in proportion to living, insulin-staining beta cells in pancreatic biopsies | 2 weeks after inclusion
Prevalence of virus infected islets in pancreatic biopsies | 2 weeks after inclusion

SECONDARY OUTCOMES:
Residual insulin secretion (C-peptide) measured by Mixed Meal Tolerance Test | 36 months after diagnosis
  Will be measured at 0, 1, 3, 9, 18, 24 and 36 months after diagnosis, but time frame is at 36 months
Insulin dosage/kilo bodyweight/24 hours | 36 months after diagnosis
  Will be calculated at 0, 1, 3, 9, 18, 24 and 36 months after diagnosis, but time frame is 36 months after diagnosis
Glycosylated hemoglobin A1 (HbA1c) | 36 months after diagnosis
  Will be measrured at 0, 1, 3, 9, 18, 24 and 36 months after diagnosis, but time frame is at 36 months. To investigate wether an eventual better endogenous insulin production gives better metabolic control, estimated by lower HbAic

CONTACTS AND LOCATIONS:
Overall Officials: Knut Dahl-Jorgensen, Prof, Principal Investigator — Oslo University Hospital
Locations (1):
- Endokrinologisk poliklinikk, Oslo Universitetssykehus Aker, Oslo, Norway